CLINICAL TRIAL: NCT02435160
Title: The Study of Efficacy and Mechanism in Fecal Microbiota Transplantation in the Treatment of Ulcerative Colitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Liu (Other)
Responsible Party: Sponsor-Investigator, Jun Liu, Shanghai general hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150406
Record Dates: First submitted 2015-04-23; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Ulcerative Colitis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

ARMS (1):
- Ulcerative Colitis (Experimental)
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation

SUMMARY:
The aim of our study is to investigate the efficacy and mechanism in fecal microbiota transplantation in the treatment of ulcerative colitis. About 20 Ulcerative Colitis (UC) patients will be recruited into our trial for Fecal Microbiota Transplantation (FMT) treatment,the safety and efficacy of FMT will be observed.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate UC patients
* male
* volunteered to our FMT trial

Exclusion Criteria:

* severe UC
* Hb < 6g/dL

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change of mayo criteria in UC patients after FMT. | one year
Number of patients with adverse events after FMT. | one year

REFERENCES:
- [Derived] Huang C, Huang Z, Ding L, Fu Y, Fan J, Mei Q, Lou L, Wang J, Yin N, Lu Y, Guo S, Zeng Y. Fecal microbiota transplantation versus glucocorticoids for the induction of remission in mild to moderate ulcerative colitis. J Transl Med. 2022 Aug 12;20(1):354. doi: 10.1186/s12967-022-03569-3. PMID 35962454